CLINICAL TRIAL: NCT02900417
Title: Evaluation of the Effect of Sitagliptin on Gut Microbiota in Patients With Newly Diagnosed Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Ji Hu, MD.,PhD., Second Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SecondSoochowU
Record Dates: First submitted 2016-08-30; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; gut microbiota; sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sitagliptin (Experimental): All the patients will receive sitagliptin 100mg daily.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — All the patients will receive sitagliptin 100mg daily
  Other Names: Sitagliptin phosphate (Januvia; Merck)

SUMMARY:
The present study will recruit 9 newly diagnosed type 2 diabetic patient to receive sitagliptin 100mg daily for 12 weeks. The aim of this study was to investigate the composition of gut microbiota before and after the therapy of sitagliptin.

DETAILED DESCRIPTION:
The present study will included 9 newly diagnosed type 2 diabetic patient to receive sitagliptin 100mg daily for 12 weeks. These patients will receive 75g oral glucose tolerance test and fasting plasma glucose levels, lipids levels, fasting insulin levels and 2 hour post-load plasma glucose levels will be measured. Stool samples will be collected before the initiation of the use of sitagliptin. After 12 weeks, all patients will have fasting plasma glucose levels, lipids levels, fasting insulin levels tested. Stool samples will be collected again.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed type 2 diabetic patients aged between 40-70 years

Exclusion Criteria:

* Any chronic disease (other than diabetes)
* Alcohol consumption/smoking
* Pregnancy/breastfeeding
* The use of antibiotics, pro-prebiotics within 3 months
* History of intestinal surgery

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
The changes of the composition of gut microbiota before and after the use of sitagliptin | 12 weeks

SECONDARY OUTCOMES:
Changes of HbA1c levels | 12 weeks
Changes of fasting plasma glucose levels, lipids levels and insulin sensitivity | 12 weeks

IPD SHARING:
Plan to Share IPD: Undecided